CLINICAL TRIAL: NCT02392013
Title: Removing Home Hazards for Older Adults
Brief Title: Home Hazard Removal Program to Reduce Falls
Acronym: HARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: US Department of Housing and Urban Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Stark, Assisstant Professor of Neurology and Occupational Therapy, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOHHU0024-14
Record Dates: First submitted 2015-03-05; First posted 2015-03-18 (Estimated); Results first posted 2024-08-30 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Accidental Falls
Keywords: older adult falls; home hazards; home barriers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Modification Group (Experimental): A tailored home-modification (home-hazard removal) intervention delivered in the home by occupational therapists over three visits and with a booster session at six months.
  Interventions: Other: Home Modification
- Usual Care Group (No Intervention): Usual care by an Area Agency on Aging

INTERVENTIONS:
Other: Home Modification — Removal of home barriers or hazards.
  Arms: Home Modification Group

SUMMARY:
This study evaluates the effectiveness and implementation of a home-hazard removal program to reduce falls in older adults through a community program delivered through the aging services network. The investigators will conduct a hybrid effectiveness/implementation trial of 300 older adults at risk for a fall who will be randomized to a home-hazard removal program or usual care and then followed for 12 months. Investigators will look at the number of falls at 6 months and 12 months.

DETAILED DESCRIPTION:
The investigators will randomly select a sample of older adults from the large observational cohort of older adults assessed annually by an Area Agendy on Aging via the National Aging Program Information System (NAPIS). The eligibility criteria include age 65 years or older and self-report of one previous fall or more in the preceding 12 months or self-report as "worried about falling." We will conduct baseline assessments and randomize participants to receive an home hazard removal program or usual care. Outcomes (falls, fall self-efficacy) will be assessed by a blinded rater at baseline and 12 months after intervention. All assessments and study visits will occur in participants' homes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years or older and self-report of one previous fall or more in the preceding 12 months or self-report as "worried about falling."

Exclusion Criteria:

* Individuals residing in nursing homes or individuals with severe cognitive impairment who are unable to give consent to participate (as determined by a score of greater than 10 on the SBT for memory10).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 310 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Stark, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Occupational Therapy Program at Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Stark S, Keglovits M, Somerville E, Hu YL, Barker A, Sykora D, Yan Y. Home Hazard Removal to Reduce Falls Among Community-Dwelling Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2122044. doi: 10.1001/jamanetworkopen.2021.22044. PMID 34463746
- [Derived] Stark S, Somerville E, Keglovits M, Conte J, Li M, Hu YL, Yan Y. Protocol for the home hazards removal program (HARP) study: a pragmatic, randomized clinical trial and implementation study. BMC Geriatr. 2017 Apr 20;17(1):90. doi: 10.1186/s12877-017-0478-4. PMID 28427336

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events occurred after participant enrollment but prior to randomization.
Period: Allocation
Arm/Group | Home Modification Group | Usual Care Group
Started | 155 | 155
Completed | 140 | 143
Not Completed | 15 | 12
Period: Follow-up
Arm/Group | Home Modification Group | Usual Care Group
Started | 140 | 143
Completed | 127 | 126
Not Completed | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Modification Group | Usual Care Group | Total
Number analyzed (Participants) | 155 | 155 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (7.7) | 74.7 (7.4) | 75 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 122 | 244
  Male | 33 | 33 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 83 | 87 | 170
  White | 72 | 67 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 155 | 155 | 310
Marital Status [Count of Participants; unit: Participants] — Population: Note. Some variables had a small amount of missing data because the participant refused a response.
  Participants
    number analyzed (Participants) | 151 | 148 | 299
    Single | 24 | 27 | 51
    Married/Partner | 29 | 30 | 59
    Divorced | 35 | 38 | 73
    Separated | 3 | 0 | 3
    Widowed | 60 | 53 | 113
Years of Education [Mean (Standard Deviation); unit: years] — Population: Note. Some variables had a small amount of missing data because the participant refused a response.
  years
    number analyzed (Participants) | 150 | 139 | 289
    (all) | 13.6 (2.8) | 13.5 (3.5) | 13.6 (3.1)
Living Status [Count of Participants; unit: Participants]
  Alone | 44 | 40 | 84
  With someone | 111 | 115 | 226
Previous Falls [Mean (Standard Deviation); unit: falls] | 1.6 (2.4) | 1.8 (4.9) | 1.7 (3.8)
Falls behavior [Mean (Standard Deviation); unit: units on a scale] — Fall prevention behavior was measured using the Falls Behavioral (FaB) Scale for the Older Person. This scale assesses the practice of 30 behaviors that could protect against falling. Response options are 1 (never), 2 (sometimes), 3 (often), and 4 (always). The average score across items is calculated, with higher scored indicating safer behaviors.
  units on a scale | 2.8 (.4) | 2.8 (.4) | 2.8 (.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Falls
Description: Prospective daily reporting of falls using a calendar
Time Frame: 12 months
Population: 135 intervention participants and 140 control participants were assessed for falls. This is different from the participant flow module, which shows that 127 intervention participants and 126 control participants completed follow-up, but the numbers in the participant flow module also took into consideration completion of secondary outcome measures.
Measure: Number; unit: falls
Arm/Group | Home Modification Group | Usual Care Group
Number analyzed (Participants) | 135 | 140
falls | 201 | 316

2. Secondary Outcome: Daily Activity Performance.
Description: Participant daily activity performance will be measured by the Older Americans Resources and Services (OARS) ADL Scale. OARS = Older Americans Resources and Services scores range from 0-28 with higher scores indicating more independence in daily activities
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Modification Group | Usual Care Group
Number analyzed (Participants) | 127 | 126
score on a scale | 21.18 (4.40) | 22.10 (4.14)

3. Secondary Outcome: Fear of Falling
Description: Concern about falling was measured using the Short Falls Efficacy Scale-International (FES-I). Respondents rate their level of concern about falling when they perform 7 different activities. Response options range from 1 (not at all concerned) to 4 (very concerned) . Scores are summed across items, and total scores range from 7 (no concern) to 28 (severe concern).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Modification Group | Usual Care Group
Number analyzed (Participants) | 127 | 126
score on a scale | 14.96 (6.23) | 14.59 (5.93)

4. Secondary Outcome: Health-related Quality of Life.
Description: Participant self-reported health will be measured using the SF-36. Patients rate responses that are then scored and transformed to a 0-100 scale where higher scores indicate greater quality of life.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Modification Group | Usual Care Group
Number analyzed (Participants) | 127 | 126
score on a scale | 42.26 (11.01) | 43.74 (11.10)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Home Modification Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 4/155 | 6/155
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/155
Other Adverse Events (participants affected / at risk) | 0/155 | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02392013/Prot_SAP_000.pdf